CLINICAL TRIAL: NCT02923895
Title: A Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: To Investigate the Efficacy of an Occluding Dentifrice in Dentinal Hypersensitivity (DH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207211
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Test dentifrice (Experimental): Participants will be instructed to dose a dry toothbrush with a full strip of toothpaste. Participants will then first brush each of the qualifying test teeth for 30 seconds each followed by the whole mouth thoroughly for at least 1 timed minute twice daily.
  Interventions: Other: Stannous fluoride
- Control dentifrice (Active Comparator): Participants will be instructed to dose a dry toothbrush with a full strip of toothpaste. Participants will brush the whole mouth thoroughly for at least 1 minute twice daily.
  Interventions: Other: Sodium monofluorophosphate

INTERVENTIONS:
Other: Stannous fluoride — 0.454% weight by weight (w/w) stannous fluoride containing 1100 parts per million (ppm) fluoride
  Arms: Test dentifrice
Other: Sodium monofluorophosphate — 0.76% w/w sodium monofluorophosphate containing 1000 ppm fluoride
  Arms: Control dentifrice

SUMMARY:
This single centre study will be used to investigate the efficacy of an experimental stannous fluoride containing dentifrice in relieving dentinal hypersensitivity (DH) after short term use compared with a standard fluoride dentifrice.

DETAILED DESCRIPTION:
This will be a single centre, three day, randomised, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), controlled study, in participants with at least two sensitive teeth that meet all the criteria at the screening and baseline (pre-treatment) visits. DH will be assessed at baseline (pre-treatment), post-treatment and after 3 days twice daily use.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged 18-65 years.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities of medical history or oral examination and absence of any condition that would impact on the participants safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* At Visit 1 (Screening): Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years; Minimum of 20 natural teeth; Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR), tooth with MGI score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1, tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response)
* At Visit 2, Baseline (Pre-treatment): Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria: Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2)

Exclusion Criteria:

* A woman who is known to be pregnant or who are intending to become pregnant over the duration of the study.
* A woman who is breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit, previous participation in this study and any participant who was randomised for inclusion in study 205710
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes and any condition which, in the opinion of the investigator, causes xerostomia.
* Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing, desensitizing treatment within 8 weeks of Screening (professional sensitivity treatments and non-dentifrice sensitivity treatments), Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of screening and vital teeth bleaching within 8 weeks of Screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening, tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, dental implants, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine and sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients).
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering andanti-inflammatory drugs, currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline and daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Creeth J, Gallob J, Sufi F, Qaqish J, Gomez-Pereira P, Budhawant C, Goyal C. Randomised clinical studies investigating immediate and short-term efficacy of an occluding toothpaste in providing dentine hypersensitivity relief. BMC Oral Health. 2019 Jun 4;19(1):98. doi: 10.1186/s12903-019-0781-x. PMID 31164116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single clinical site in Canada.
Pre-assignment Details: A total of 197 participants were screened and enrolled in the study, out of which 192 participants were randomized to the study treatments. Five participants were not randomized: 1 participant was screening failure, and 4 participants withdrew their consent.
Groups:
- Test Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of toothpaste. Participants then first brushed each of the qualifying test teeth for 30 seconds each followed by the whole mouth thoroughly for at least 1 timed minute twice daily.
- Control Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of toothpaste. Participants brushed the whole mouth thoroughly for at least 1 minute twice daily.
Period: Overall Study
Arm/Group | Test Dentifrice | Control Dentifrice
Started | 97 | 95
Completed | 97 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice | Control Dentifrice | Total
Number analyzed (Participants) | 97 | 95 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (12.95) | 46.9 (10.53) | 46.9 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 72 | 140
  Male | 29 | 23 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 12 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 31 | 49
  White | 62 | 51 | 113
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 3
Description: The examiner assessed the participant's response to an evaporative air stimulus for each of the two test tooth using the Schiff Sensitivity Scale which was scored as follows: 0 Participant does not respond to air stimulation, 1 Participant responds to air stimulus but does not request discontinuation of stimulus, 2 Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3 Participant responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. The Schiff sensitivity score was calculated as the average of individual test teeth score. Change from baseline in Schiff sensitivity was calculated as participant level mean change from baseline of the 2 test teeth. A reduction in Schiff Sensitivity score was indicative of an improvement in sensitivity.
Time Frame: Baseline and Day 3
Population: Analysis for this outcome was performed on Intent-to-treat (ITT) population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 97 | 95
Score on a scale
  At Baseline (Day 0, Pre-treatment) | 2.44 (0.450) | 2.49 (0.475)
  At Day 3 | 1.01 (0.956) | 2.37 (0.571)
  Change from Baseline | -1.44 (0.811) | -0.13 (0.431)
Statistical Analysis 1: Comparison: Test Dentifrice vs Control Dentifrice; Test type: Superiority — All statistical analyses were conducted under the null hypothesis (H0) of no difference between treatments versus the alternate hypothesis (H1) of a difference between treatments; p < .0001, ANCOVA — From ANCOVA model with change from baseline in Schiff Sensitivity Score as response and treatment as a factor and baseline Schiff sensitivity score as a covariate; Mean Difference (Net) = -1.31, 95% CI 2-sided [-1.500 to -1.128] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Tactile Threshold on Day 3
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 gram[g] to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline and Day 3
Population: Analysis for this outcome was performed on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 97 | 95
g
  At Baseline | 13.40 (4.242) | 13.58 (4.416)
  At Day 3 | 39.28 (20.979) | 14.89 (6.357)
  Change from Baseline | 25.88 (19.804) | 1.32 (6.111)

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score After a Single Use
Description: as for outcome 1
Time Frame: Baseline to 60 seconds post first treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 97 | 95
Score on a scale
  At Baseline (Day 0, Pre-treatment) | 2.44 (0.450) | 2.49 (0.475)
  Day 0 (Post-treatment) | 1.76 (0.781) | 2.40 (0.534)
  Change from Baseline | -0.68 (0.704) | -0.09 (0.401)

4. Secondary Outcome: Change From Baseline in Tactile Threshold After a Single Use
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline to 60 seconds post first treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 97 | 95
g
  At Baseline (Day 0, Pre-treatment) | 13.40 (4.242) | 13.58 (4.416)
  Day 0, Post-treatment | 22.47 (11.839) | 14.63 (6.069)
  Change from Baseline | 9.07 (11.418) | 1.05 (5.644)

ADVERSE EVENTS:
Time Frame: Approximately 64 days (from Screening Visit to till 5 days following last administration of study product on Visit 3)
Groups:
- Control Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of toothpaste. Participants then brushed the whole mouth thoroughly for at least 1 minute twice daily.
Arm/Group | Test Dentifrice | Control Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/95
Other Adverse Events (participants affected / at risk) | 1/97 | 0/95
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=97) | Control Dentifrice (N=95)
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.